CLINICAL TRIAL: NCT00854945
Title: A Phase 1/2, Single-Arm Study To Assess The Efficacy and Safety Of 72-Hour Continuous Intravenous Dosing Of ON 01910.Na Administered Every Other Week in Patients With Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML)
Brief Title: Study of 72-Hour Infusion of ON 01910.Na in Patients With MDS or AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-15
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Myelodysplastic Syndrome; Refractory Cytopenia; Refractory Anemia; Dysplasia; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Cytopenia; Anemia, Refractory | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ON 01910.Na (Experimental): 1800 mg/day of ON 01910.Na administered as a 24-hour continuous intravenous infusion on days 1, 2 and 3 of 14-day cycle.
  Interventions: Drug: ON 01910.Na

INTERVENTIONS:
Drug: ON 01910.Na — 1800 mg/day as a 24-hour continuous intravenous infusion administered three times a week every 2 weeks
  Other Names: ON 01910; rigosertib

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of ON 01910.Na Concentrate when it is administered as an intravenous continuous infusion (IVCI) over 72 hours once every 2 weeks in a broad population of MDS patients. Rationale for this study is based on the activity observed in another study with ON 01910.Na in patients with refractory anemia with excess blasts (RAEB) 1 and 2 MDS. This study will examine ON 01910.Na in a broader population of MDS and AML patients. This phase I/II study will establish the Maximum Tolerated Dose (MTD) starting with a dose of 800 mg/m2 per day administered over 24 hours for 2 consecutive days as a continuous intravenous infusion, once a week for 3 weeks of a 4-week cycle and examine the efficacy and safety profile at the MTD.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of ON 01910.Na CIV 24-hour infusion administered three times a week every other week in achieving by week 25 a complete or partial response as defined per the 2000 International Working Group (IWG) Criteria in patients with MDS or as defined by Cheson et al. [JCO 21:4642 (2003)] in patients with AML.

The secondary objectives are to assess:

* Time and duration of response
* Blastic response in bone marrow
* Improvement of dyspoiesis as evaluated by the change in aneuploidy in bone marrow
* Change in International Prognostic Scoring System (IPSS) in MDS patients
* Major and minor responses in absolute neutrophil count, according to IWG 2000 criteria
* Major and minor responses in platelet count, according to IWG 2000 criteria
* Major and minor erythroid response, according to IWG 2000 criteria
* Time to progression
* Overall survival at 25 and 50 weeks
* Proportion of MDS patients transitioning to acute myeloid leukemia (AML) at 25 and 50 weeks

This is a phase 1/2 single arm study in which six to thirty-five patients with MDS or AML who meet all other inclusion/exclusion criteria will receive ON 01910.Na as an intravenous continuous infusion (IVCI) over 72 hours once a week every other week.

In the phase 1 portion of the study, a traditional dose escalation rule, also known as the "3+3" rule, will be used. Three patients will be treated at the 800 mg/m2/day dose level. If none of the patients experience a DLT during cycle 1, the next group of 3 patients will receive 1500 mg/m2/day. If no DLT is seen at the 1500 mg/m2/day dose level, then the dose used in the phase 2 portion of the study will be 1500 mg/m2/day. If there is DLT in one of the first three patients at the 800 mg/m2/day dose level, this dose level will be expanded to 6 patients. If ≤ 1 patient out of 6 experience DLT, then the dose will be escalated to the 1500 mg/m2/day dose level. If ≥ 2 patients experience DLT at the 800 mg/m2/day dose level, a full safety review will determine if further enrollment of patients will proceed. If there is DLT in one of the first three patients at the 1500 mg/m2/day dose level, this dose level will be expanded to 6 patients. If ≤ 1 patient out of 6 experience DLT at the 1500 mg/m2/day dose level, then 1500 mg/m2/day dose level will be considered the MTD. If ≥ 2 patients experience DLT at the 1500 mg/m2/day dose level, then 800 mg/m2/day will be designated as the MTD.

The total study duration is 29 weeks, which includes a 2-week screening phase, a 23-week dosing phase, and a 4-week follow-up phase that begins after the last dose of ON 01910.Na. Beginning at week 4, and every 2 weeks thereafter, patients will be assessed for response and followed up.

Patients who achieve by week 25 a complete or partial response or stabilization of their disease are eligible to receive an additional 24 weeks of ON 01910.Na 1800 mg/24 h for 72 h once a week every 2 weeks and will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Diagnosis of MDS or AML via bone marrow aspirate and biopsy performed within 8 weeks prior to study entry according to WHO Criteria and FAB Classification. AML patients must be:

not eligible for standard chemotherapy, including newly diagnosed patients over 70 years; with relapsed or refractory AML; and, with AML secondary to prior cancer chemotherapy or evolving from a myeloproliferative/myelodysplastic syndrome.

* Anemia requiring transfusion support with at least one unit of packed red blood cells per month for greater than or equal to 2 months or Hemoglobin < 10 g/dL OR Thrombocytopenia (platelet count < 100,000/µl) OR Neutropenia (absolute neutrophil count < 1,500/µl)
* Failed to respond to, relapsed following, or opted not to participate in bone marrow transplantation
* Off all other treatments for MDS or AML (including filgrastim (G-CSF) and erythropoietin) for at least four weeks. As an exception, filgrastim (G-CSF) can be used before, during and after the protocol treatment for patients with documented febrile neutropenia (<500/µl)
* ECOG Performance Status 0, 1 or 2
* Adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study for female patients of reproductive potential
* Female patient with reproductive potential must have a negative serum beta-HCG pregnancy test at screening
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Patient (or his/her legally authorized representative) must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Anemia due to factors other than MDS or AML (including hemolysis or gastrointestinal bleeding)
* Proliferative (WBC ≥ 12,000/mm3) chronic myelomonocytic leukemia
* Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* History of HIV-1 seropositivity
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin > 1.5 mg/dL not related to hemolysis or Gilbert's disease, ALT or AST > 2 X ULN
* Serum creatinine > 1.5 mg/dL or calculated creatinine clearance < 60 ml/min/1.73 m2
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <134 Meq/L).
* Women patients who are pregnant or lactating
* Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Uncontrolled hypertension (defined as a systolic pressure ≥ 160 and/or a diastolic pressure ≥ 110)
* New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures
* Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Response as defined per the 2000 International Working Group (IWG) Criteria in patients with MDS. | 6 -12 months

SECONDARY OUTCOMES:
Hematologic improvement. | 6 - 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Azra Raza, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Background] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Result] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.